CLINICAL TRIAL: NCT00440401
Title: A Randomised, Open Label, Parallel-group, Multi-centre Trial to Compare the Efficacy and Safety of TachoSil® Versus Standard Haemostatic Treatment in Cardiovascular Surgery
Brief Title: TachoSil® Versus Standard Haemostatic Treatment of Haemorrhage in Cardiovascular Surgery (TC-023-IM)
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Nycomed (Industry)
Responsible Party: Nycomed, Clinical Trial Operations
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: TC-023-IM
Record Dates: First submitted 2007-02-26; First posted 2007-02-27 (Estimated); Results first posted 2010-06-04 (Estimated); Last update posted 2012-05-08 (Estimated); Status verified 2010-07

CONDITIONS: Haemorrhage; Haemostasis; Cardiovascular Surgery
Keywords: Surgical treatment of haemorrhage
MeSH Terms: conditions — Hemorrhage | interventions — Fibrinogen; Thrombin; Cardiovascular Surgical Procedures

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- TachoSil® (Active Comparator)
  Interventions: Drug: fibrinogen (human) + thrombin (human)
- Standard Treatment (Active Comparator): Standard Treatment of haemorrhage in cardiovascular surgery
  Interventions: Drug: Standard haemostatic treatment in cardiovascular surgery

INTERVENTIONS:
Drug: fibrinogen (human) + thrombin (human)
  Arms: TachoSil®
Drug: Standard haemostatic treatment in cardiovascular surgery — Any haemostatic fleece material without additional active coagulation stimulating compounds (primarily Surgicel®)
  Arms: Standard Treatment

SUMMARY:
To demonstrate efficacy and safety of TachoSil® in cardiovascular surgery

ELIGIBILITY:
Inclusion Criteria:

All inclusion criteria must be answered "yes" for a subject to participate in the trial.

At Screening:

1. Has the subject given informed consent according to local requirements before any trial related activities? A trial related activity is any procedure that would not have been performed during the routine management of the subject. In this trial the screening is the first trial related activity.
2. For female subjects of childbearing potential: Is the pregnancy test at screening negative?
3. Does the female subject of childbearing potential use adequate contraception (contraceptive pill, contraceptive injection, contraceptive implant or intrauterine device)?
4. Is the subject ≥ 18 years of age?
5. Is the following planned: An elective surgery on the heart, the ascending aorta or arch, requiring cardiopulmonary bypass procedure?

   Intra operative (after primary haemostatic treatment):
6. Is bleeding from the heart muscle, the pericardium, a major vessel or a vascular bed that requires supportive haemostatic treatment present?
7. Has the area with the most problematic haemorrhage (target area) been identified? (please note that this must be done before randomisation).
8. Is it possible to compress the randomised treatment (TachoSil® or control fleece material) for 3 minutes?

Exclusion Criteria:

All exclusion criteria must be answered "no" for a subject to participate in the trial.

At Screening:

1. Has the subject participated in any other trial with an investigational drug or device within 30 days before inclusion in this trial?
2. Does the subject participate in a clinical trial concomitantly with the present trial?
3. Is the subject undergoing an emergency operation?
4. Has the subject a history of allergic reactions after application of human fibrinogen, human thrombin and/or collagen of any origin?
5. Is the subject suffering from known coagulopathy?
6. Is the subject currently participating or has the subject previously participated in the TC-023-IM trial?
7. Is the female subject pregnant or breast feeding?

   Intra operative (after primary haemostatic treatment):
8. Has liquid fibrin sealant/glue or TachoSil® been applied?
9. Has the following occurred: Disseminated intravascular coagulation (DIC), i.e. micro vascular bleeding?

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2007-02; Primary Completion 2007-08 (Actual); Study Completion 2007-11 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Nycomed Clinical Trial Operations, Study Chair — Headquaters
Locations (1):
- Nycomed, Roskilde, Denmark

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: From the total of 120 enrolled subjects, data are presented for 119 randomised subjects that received trial treatment (= Intention to Treat (ITT) population).
Groups:
- TachoSil®: Absorbable sponge for intra-operative topical application
- Comparator: Standard haemostatic treatment in cardiovascular surgery
Period: Overall Study
Arm/Group | TachoSil® | Comparator
Started | 59 | 60
Completed | 55 | 54
Not Completed | 4 | 6
Not completed — Adverse Event | 2 | 1
Not completed — Other | 2 | 5

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | TachoSil® | Standard Treatment | Total
Number analyzed (Participants) | 59 | 60 | 119
Age, Customized [Number; unit: participants]
  18-65 years | 24 | 21 | 45
  65 years or above | 35 | 39 | 74
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 14 | 17 | 31
  Male | 45 | 43 | 88
Race/Ethnicity, Customized [Number; unit: participants] — All patients were Caucasian
  participants
    Caucasian | 59 | 60 | 119
Classification of surgery [Number; unit: Percentage of subjects] — Planned elective surgery on the heart, the ascending aorta or arch, requiring cardiopulmonary bypass procedure.
  The information about planned surgery reflects the protocol defined eligibility criterion no. 5. In addition, the actually performed surgery is categorized into simple and combined/complex cardiovascular procedures. The proportions of patients undergoing combined/complex cardiovascular procedures in the TachoSil® group and the Standard Treatment group, respectively, were 44 and 59 percent. The calculated total (103) is irrelevant and inappropriate arithmetic.
  Percentage of subjects | 44 | 59 | 103
Evaluation of bleeding at target area before randomization [Number; unit: participants] — In order to avoid selection bias, evaluation of bleeding at target area was performed after completion of primary hemostasis and prior to randomization.
  Data obtained prior to final assessment of patient eligibility and randomization.
  More than one record/condition per patient possible.
  participants
    Arterial | 48 | 40 | 88
    Venous | 11 | 20 | 31
    Mild haemorrhage | 19 | 24 | 43
    Moderate haemorrhage | 35 | 34 | 69
    Severe haemorrhage | 5 | 2 | 7
Identification of target area for efficacy evaluation [Number; unit: participants] — In order to avoid selection bias, intra-operative randomization was only performed if supportive haemostatic treatment was required after completion of primary haemostasis.
  Data obtained prior to final assessment of patient eligibility and randomization.
  More than one record/condition per patient possible.
  participants
    Aorta | 35 | 32 | 67
    Coronary anastomosis | 2 | 3 | 5
    Internal mammary artery vascular bed | 1 | 1 | 2
    Left atrium | 3 | 2 | 5
    Left ventricle | 3 | 2 | 5
    Right atrium | 5 | 10 | 15
    Right ventricle | 11 | 8 | 19
    Other | 3 | 2 | 5
Primary haemostatic treatment [Number; unit: participants] — Data obtained prior to final assessment of patient eligibility and randomization.
  More than one record/condition per patient possible.
  participants
    Suturing | 43 | 43 | 86
    Electro-coagulation | 6 | 5 | 11
    Clips | 3 | 2 | 5
    Gauze | 0 | 1 | 1
    None | 10 | 12 | 22
Type of tissue [Number; unit: participants] — Type of tissue treated with randomized treatment
  participants
    Tissue | 16 | 22 | 38
    Vessel | 43 | 38 | 81

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Subjects Achieving Haemostasis at 3 Minutes
Description: Three minutes after application of trial treatment (TachoSil® or standard fleece material) the investigator evaluated if haemostasis in the target area was achieved.
Time Frame: 3 minutes
Population: Three subjects were randomised to standard treatment but incorrectly received TachoSil® instead. All other subjects received the trial treatment to which they were randomised. The intention to treat (ITT) population was defined "as randomised" and the Safety population (= basis for Adverse Events analyses) was defined "as treated".
Measure: Number (95% Confidence Interval); unit: Proportion of Subjects
Arm/Group | TachoSil® | Standard Treatment
Number analyzed (Participants) | 59 | 60
Proportion of Subjects | 0.746 [0.635 to 0.857] | 0.333 [0.214 to 0.453]
Statistical Analysis 1: Comparison: TachoSil® vs Standard Treatment; Test type: Superiority or Other; p < 0.0001, Cochran-Mantel-Haenszel; Normal approximation to the binominal distribution is used to construct the asymptotic confidence intervals

2. Secondary Outcome: Proportion of Subjects Achieving Haemostasis at 6 Minutes.
Description: Six minutes after application of trial treatment (TachoSil® or standard fleece material) the investigator evaluated if haemostasis in the target area was achieved.
Time Frame: 6 minutes
Population: as for outcome 1
Measure: Number (95% Confidence Interval); unit: Proportion of Subjects
Arm/Group | TachoSil® | Standard Treatment
Number analyzed (Participants) | 59 | 60
Proportion of Subjects | 0.949 [0.893 to 1.000] | 0.717 [0.603 to 0.831]
Statistical Analysis 1: Comparison: TachoSil® vs Standard Treatment; Test type: Superiority or Other; p < 0.0006, Cochran-Mantel-Haenszel; Normal approximation to the binominal distribution is used to construct the asymptotic confidence intervals

ADVERSE EVENTS:
Description: SAE/AE assessment by neutral questioning "Have you experienced any health problems since the last contact?" by the investigator at each contact (visit or phone).
  Basis for analysis was the safety population (= all subjects randomised and given trial treatment).
Arm/Group | TachoSil® | Standard Treatment
Serious Adverse Events (participants affected / at risk) | 8/62 | 18/57
Other Adverse Events (participants affected / at risk) | 38/62 | 30/57
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TachoSil® (N=62) | Standard Treatment (N=57)
Atrial fibrillation (Cardiac disorders) | 1 (1) | 4 (4)
Atrioventricular block third degree (Cardiac disorders) | 0 (0) | 4 (4)
Cardiac arrest (Cardiac disorders) | 0 (0) | 1 (1)
Cardiac tamponade (Cardiac disorders) | 1 (2) | 1 (1)
Low cardiac output syndrome (Cardiac disorders) | 0 (0) | 2 (2)
Myocardial infarction (Cardiac disorders) | 0 (0) | 2 (2)
Ventricular tachycardia (Cardiac disorders) | 0 (0) | 2 (2)
Colitis ischaemic (Gastrointestinal disorders) | 0 (0) | 1 (1)
Multi-organ failure (General disorders) | 2 (2) | 1 (1)
Mediastinitis (Infections and infestations) | 1 (1) | 0 (0)
Pneumonia klebsiella (Infections and infestations) | 0 (0) | 1 (1)
Postoperative wound infection (Infections and infestations) | 0 (0) | 1 (1)
Sepsis (Infections and infestations) | 0 (0) | 2 (2)
Staphylococcal bacteraemia (Infections and infestations) | 1 (1) | 0 (0)
Wound infection (Infections and infestations) | 2 (2) | 0 (0)
Wound infection staphylococcal (Infections and infestations) | 1 (1) | 0 (0)
Brain contusion (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cardiac function disturbance postoperative (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Haemothorax (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 (1) | 0 (0)
Post procedural stroke (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Stent-graft endoleak (Injury, poisoning and procedural complications) | 0 (0) | 1 (1)
Cerebral infarction (Nervous system disorders) | 1 (1) | 0 (0)
Cerebrovascular accident (Nervous system disorders) | 0 (0) | 1 (1)
Vocal cord paralysis (Nervous system disorders) | 0 (0) | 1 (1)
Mental disorder due to a general medical condition (Psychiatric disorders) | 0 (0) | 1 (1)
Renal failure acute (Renal and urinary disorders) | 1 (1) | 1 (1)
Tubulointerstitial nephritis (Renal and urinary disorders) | 1 (1) | 1 (1)
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (5)
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 2 (2)
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1)
Haemorrhage (Vascular disorders) | 0 (0) | 1 (1)
Hypotension (Vascular disorders) | 0 (0) | 1 (1)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | TachoSil® (N=62) | Standard Treatment (N=57)
Haemorrhagic anaemia (Blood and lymphatic system disorders) | 5 (5) | 6 (6)
Atrial fibrillation (Cardiac disorders) | 17 (17) | 10 (10) — non-serious
Bradycardia (Cardiac disorders) | 1 (1) | 3 (3)
Pericardial effusion (Cardiac disorders) | 3 (3) | 4 (4)
Tachyarrhythmia (Cardiac disorders) | 4 (4) | 4 (4)
Constipation (Gastrointestinal disorders) | 3 (3) | 3 (3)
Nausea (Gastrointestinal disorders) | 8 (8) | 5 (5)
Pyrexia (General disorders) | 4 (4) | 3 (3)
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 2 (2) | 3 (3) — non-serious
Haemoglobin decreased (Investigations) | 0 (0) | 3 (3)
Hyperglycaemia (Metabolism and nutrition disorders) | 6 (6) | 7 (7)
Psychotic disorder (Psychiatric disorders) | 0 (0) | 4 (4)
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 14 (14) | 9 (9) — non-serious
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 4 (4) | 2 (3)
Hypotension (Vascular disorders) | 2 (2) | 4 (4) — non-serious

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less